CLINICAL TRIAL: NCT01022294
Title: Analgetic Effect of Nitrousoxide-oxygen Inhalation for Dental Treatment of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: M-20070261
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Dental Pain; Muscle Sensitivity to Pressure; Skin Sensitivity to Electric Stimulation
Keywords: children; analgesia; dental treatment; inhalation
MeSH Terms: conditions — Toothache; Agnosia; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Inhalation of nitrousoxide-oxygen during the first experimental session; inhalation of atmospheric air during the second session
  Interventions: Drug: Nitrousoxide-oxygen and atmospheric air
- Arm 2 (Experimental): Inhalation of atmospheric air during the first experimental session; inhalation of nitrousoxide-oxygen during the second session
  Interventions: Drug: Atmospheric air; nitrousoxide-oxygen

INTERVENTIONS:
Drug: Nitrousoxide-oxygen and atmospheric air — Nitrousoxide-oxygen and atmospheric air
  Other Names: Nitrousoxide-oxygen first
  Arms: Arm 1
Drug: Atmospheric air; nitrousoxide-oxygen — Atmospheric air; nitrousoxide-oxygen
  Other Names: Atmospheric air first
  Arms: Arm 2

SUMMARY:
To assess the analgetic effect of nitrousoxide-oxygen inhalation on pain perception in 12-15 years old children from 1) the dental pulp; 2) the masseter muscle; 3) the skin on the upper lip

DETAILED DESCRIPTION:
The present study is a randomized, cross-over blinded study on the analgetic effect of nitrousoxide-oxygen on sensitivity of the dental pulp, the skin and muscles.

It is conducted in healthy 12-15 year old Danish children attending public schools in the municipality of Aarhus, Denmark

ELIGIBILITY:
Inclusion Criteria:

* ASA-groups I or II
* 12-15 year of age
* sound upper central incisors

Exclusion Criteria:

* difficulties breathing through the nose
* pregnancy
* trauma to test teeth

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Dental pain (pulp) threshold | During and after inhalation

SECONDARY OUTCOMES:
Muscle sensitivity to pressure | During and after inhalation
Skin sensitivity ot electric stimulation | During and after inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poulsen, dr.odont., Study Chair — Dept. of Pediatric Dentsitry, School of Dentistry, Faculty of Health Sciences, Aarhus University, Denmark
Locations (1):
- Dept. of Pediatric Dentistry, School of Dentistry, Faculty of Health Sciences, Aarhus University, Aarhus, Denmark